CLINICAL TRIAL: NCT00711815
Title: Biomarkers of HPV Clearance: A Prospective Study
Brief Title: A Study to Identify Markers in Blood and Tissue of HPV Clearance
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Warner K. Huh, M.D., UAB
Other Study IDs: W061101002 (UAB 0626); 20062154 (WIRB); T06020012
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: HPV Infections
Keywords: Women of the state of Alabama; CIN 1; negative biopsy; normal colposcopy; HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, cervical cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- UA: HPV positive

SUMMARY:
This is a research study looking at gene characteristics in blood and Pap smear samples in hopes of identifying markers that will predict if the HPV infection is present or not.

DETAILED DESCRIPTION:
Because infection with high-risk human papillomavirus is a necessary cause of cervical cancer, HPV testing has many potential uses in cervical cancer screening. Unfortunately, like cytology, it suffers from a lack of specificity when used for population-based screening. Given that HPV testing detects more cases of CIN3+ than cytology and that it would probably be more practical in developing regions, finding a biomarker that would increase specificity has been the goal for much research on HPV and cervical cancer. The goal of this study is to explore potential predictors of viral clearance, specifically RNA levels of candidate genes in cervical swabs and host genetic polymorphisms, in the context of genotype-specific infection data.

ELIGIBILITY:
Inclusion Criteria:

* HPV positive

Exclusion Criteria:

* Negative for HPV

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HPV-positive women with biopsy-confirmed CIN 1 or negative biopsies or normal colposcopic findings
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2007-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warner K Huh, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States